CLINICAL TRIAL: NCT02681705
Title: Phase 2 Study of Radiation Therapy and Combination Chemotherapy Following Surgery in Treating Children With Newly Diagnosed Medulloblastoma
Brief Title: Radiation Therapy and Combination Chemotherapy for Medulloblastoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Chuanying Zhu, doctor, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: sanghaixinhua-003
Record Dates: First submitted 2016-02-10; First posted 2016-02-12 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Medulloblastoma
MeSH Terms: conditions — Medulloblastoma | interventions — Temozolomide; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study Treatment (Experimental): All subjects will undergo routine surgical staging of their tumor. Treatment must begin within 28 days of surgery. Craniospinal Radiation therapy will last for 6 weeks, five days per week. Once a week during radiation, subjects will also be treated with Temozolomide. Temozolomide is applied to these patients as a chemotherapy drug with a dosage of 75mg/m2, daily. The chemotherapy and radiation therapy are combined as Temozolomide is taken 1 hour prior to every fraction of radiotherapy. In 4 weeks after the completion of radiotherapy, temozolomide is given for 8 cycles.
  Interventions: Drug: Temozolomide; Radiation: Craniospinal Radiation

INTERVENTIONS:
Drug: Temozolomide — Temozolomide is applied to these patients as a chemotherapy drug with a dosage of 75mg/m2, daily. The chemotherapy and radiation are combined as temozolomide is taken 1 hour prior to every fraction of radiotherapy. In 4 weeks after the completion of radiotherapy, temozolomide is given for 8 cycles (dosage: the 1st cycle, 150mg/m2, daily × 5 days, 4 weeks a cycle; the 2-8th cycle, 200mg/m2, daily × 5 days, 4 weeks a cycle and repeated again).
  Other Names: brand names Temodar and Temodal and Temcad
Radiation: Craniospinal Radiation — Craniospinal radiation will begin within 28 days of surgery. Craniospinal Radiation therapy will last for 6 weeks, five days per week. Once a week during radiation, subjects will also be treated with chemotherapy (Temozolomide).
  Other Names: Radiation

SUMMARY:
This phase II trial is studying giving radiation therapy together with combination chemotherapy after surgery to see how well it works in treating children with newly diagnosed medulloblastoma.

DETAILED DESCRIPTION:
OUTLINE:

Adjuvant induction chemoradiotherapy: Beginning within 28 days after prior resection, patients undergo radiotherapy to the craniospinal axis 5 days a week for 4 weeks and then conformal radiotherapy to the tumor bed 5 days a week for 2 weeks. Beginning 1 week after the initiation of radiotherapy, Temozolomide is applied to these patients as a chemotherapy drug with a dosage of 75mg/m2, daily. The chemotherapy and radiation are combined as temozolomide is taken 1 hour prior to every fraction of radiotherapy.

Maintenance chemotherapy: Beginning 4 weeks after the completion of induction chemoradiotherapy, patients receive eight 4-week cycles of temozolomide (dosage: the 1st cycle, 150mg/m2, daily × 5 days, 4 weeks a cycle; the 2-8th cycle, 200mg/m2, daily × 5 days, 4 weeks a cycle and repeated again).

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed posterior fossa medulloblastoma
2. No residual tumor greater than 1.5 cm^2 after resection by postoperative MRI No tumor in the spinal or cerebral subarachnoid space by MRI No tumor in the subarachnoid space by Cerebrospinal fluid (CSF) No failure to perform staging studies (spine MRI and CSF cytology) preoperatively or postoperatively
3. Must begin radiotherapy on study within 28 days after surgery

Exclusion Criteria:

1. Prior radiotherapy and anti-tumor chemotherapy other than corticosteroids are not allowed.
2. Patients must begin radiotherapy on protocol within 28 days of completion of surgery. Exceptions need to be approved by the Principal Investigator.
3. Patients with the following will not be eligible:

> 1.5cm3 residual tumor following resection as indicated by post-operative MRI. tumor in spinal or cerebral subarachnoid space either by MRI of brain and spine tumor in subarachnoid space by CSF cytology failure to perform staging studies (spine MRI, CSF cytology) either pre- or post- operatively

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2010-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | first analysis will occur 1 month after accrual of all patients

SECONDARY OUTCOMES:
Progression free survival(PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
Overall survival (OS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
Evaluate Rate of Late Neurotoxic Effects | 3 years
  Evaluate the late neurotoxic effects of low dose craniospinal radiation, including cognitive, endocrinologic and auditory function.

CONTACTS AND LOCATIONS:
Overall Officials: mawei jiang, MD, Principal Investigator — The Department of Radiation Oncology, Xin Hua Hospital affiliated to Shanghai Jiaotong University School of Medicine
Locations (1):
- The Department of Radiation Oncology, Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes